CLINICAL TRIAL: NCT06724172
Title: CHIME: Comparing Health Interventions for Maternal Equity
Acronym: CHIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jennifer Woo Baidal, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77034; 20244792 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Overweight; Nutrition; Chronic Disease; Diabetes; Pregnancy
MeSH Terms: conditions — Obesity; Overweight; Chronic Disease; Diabetes Mellitus | interventions — Self-Management

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Management (Experimental): A self-management intervention through direct provision of social needs supports (grocery, physical activity, and transportation support) with self-directed behavior change tools and usual care.
  Interventions: Behavioral: Self-Management
- Community-Based (Experimental): A community-based intervention for active social needs referrals assistance with health coaching and active lifestyle intervention and usual care.
  Interventions: Behavioral: Community-Based
- Usual Care (No Intervention): Patients randomized to the usual care control group will not receive the study interventions. Instead, these patients will receive usual care which includes social needs screening in the clinical setting, targeted community service and program referrals, clinical decision support tools for social needs support in the electronic health record, and routine clinical care with provider-based lifestyle counseling.

INTERVENTIONS:
Behavioral: Self-Management — We will universally offer social needs supports (grocery, physical activity, transportation support) widely in use in clinical settings. Patients may elect to receive all, some, or none of the supports. The patient-directed, structured self-management intervention will be provided through mobile health technology (mHealth) and/or mailings, according to patient preference. Participants will receive health information to support health education and behavior change.
  Arms: Self-Management
Behavioral: Community-Based — As is currently in use broadly by community health workers, participants will complete a detailed social needs assessment and active assistance with referrals to evidence-based home visiting programs; maternal child health services to promote social support and resource access; and services to improve social determinants of health including active enrollment assistance for WIC, SNAP, healthcare and insurance, legal support, housing, job training, mental health and others. Community health workers will deliver group and individual physical activity support and assistance with behavioral goal setting.
  Arms: Community-Based

SUMMARY:
The goal of this comparative effectiveness trial is to compare how three different approaches to overcome barriers to resources and provide nutrition and physical activity counseling improve maternal healthy weight in pregnancy and postpartum.

The main question it aims to answer is which of the two multi-level, multi-component interventions has greater effectiveness in reducing maternal postpartum weight retention at 12-months postpartum.

Hypothesis (primary): Both multi-level, multi-component interventions will have greater effectiveness reducing maternal postpartum weight retention at 12-months postpartum than the usual care group.

Hypothesis (secondary): The community-based intervention will have greater effectiveness than the self-management intervention.

Participants will be asked to participate in one of the study interventions from early pregnancy until 12 months postpartum and complete five research visits. General procedures include completion of:

* Questionnaires
* Dietary recalls
* In-depth interviews
* Anthropometric measurements
* Collection of blood via finger stick or blood panel

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 18 years or older
* Maternal gestational age ≤ 20 weeks with viable singleton pregnancy documented on first trimester ultrasound with an intention to continue pregnancy to term
* Plans to continue receiving antenatal care at the recruitment site/network
* Maternal characteristics include at least one of the following:
* Self identifies as Black/African American
* Self identifies as Hispanic/Latino/a/e/x
* Insured by Medicaid
* Maternal ability to speak English or Spanish
* Completion of baseline data collection (maternal survey data, weight, and height measurement prior to randomization)

Exclusion Criteria:

* Age < 18 years at baseline because of unique developmental differences of adolescents and regulations regarding age of consent
* Underweight (BMI <18 kg/m2) at pre-pregnancy period
* Underlying disease/treatment that might impact weight status (e.g., significant gastrointestinal conditions, major psychiatric disorders, and others at the discretion of the study clinician)
* Unwillingness or inability to complete study visits or intervention components
* Unwillingness or inability to commit to intervention components for self or infant, including plans to move more than 100-mile radius from recruitment site
* Multiple gestations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 795 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Maternal postpartum weight retention at 12-months postpartum. | From enrollment to the end of the intervention at 12 months postpartum.
  The primary outcome will be calculated as the difference between baseline weight and 12-month postpartum weight. Baseline weight will be defined as the first clinical measure of maternal weight prior to 12 weeks gestation.

SECONDARY OUTCOMES:
Household social needs and maternal perinatal health outcomes | From enrollment to the end of the intervention at 12 months postpartum.
  We will obtain patient self-reported measures where applicable for secondary outcomes through validated questionnaires. Secondary outcomes include household food security, gestational weight gain, gestational diabetes, with maternal race and ethnicity and pre-pregnancy body mass index category as effect modifiers.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - New York Presbyterian Queens, Flushing, New York

IPD SHARING:
Plan to Share IPD: No